CLINICAL TRIAL: NCT01646099
Title: Internet-Based Sun Protection Program for Kidney Transplantation Recipients
Brief Title: Sun Protection of Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Research Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00058220
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Unspecified Complication of Kidney Transplant; Disorder Related to Renal Transplantation
Keywords: Kidney transplant; Renal transplant; Sun protection; Skin cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sun Protection Education (Experimental): Distribution of the internet-based sun protection educational program.
  Interventions: Behavioral: Internet-based sun protection education
- Control (No Intervention): Distribution of general skin care information.

INTERVENTIONS:
Behavioral: Internet-based sun protection education — Prior to summer, KTRs who agree to participate will receive a text message with their access code to the Internet intervention to access from their homes on a personal device. After online completion of baseline assessments, participants will be randomized to receive the intervention or general skin care information (control). Following the initial use, the participants may revisit the Internet intervention on a personal device or at the doctor's office on a tablet PC. Over the next 6 weeks, sun protection text reminders will be sent to intervention KTRs' cell phones and they will respond that they read the message. Control participants will receive text messages about general skin care.
  Arms: Sun Protection Education

SUMMARY:
This study is being done to evaluate the effectiveness of a Sun Protection Strategies internet-based program for kidney transplant recipients. Since the medication taken to preserve the kidney transplant puts kidney transplant recipients at increased risk of developing a sunburn as well a skin cancer, the program will help people learn how to practice effective sun protection for their condition.

DETAILED DESCRIPTION:
Cognitive interviews about an internet-based sun protection strategies program will be performed with up to 45 kidney transplant recipients (KTRs) who have participated in past surveys. A second group of 150 KTRs will be asked to evaluate the internet-based module for the effectiveness of information. A third group of 12 KTRs will be asked to evaluate the internet-based module for usability. A fourth group of 160 KTRs will be asked to take part in a randomized controlled trial evaluating the fully developed internet-based sun protection strategies program.

Kidney transplant recipients (KTRs) are at risk to develop skin cancer. Adequate sun protection after transplantation can reduce the risk of developing skin cancer. In 2006, the National Kidney Foundation (NKF) found that sun protection education delivery and content varied among transplantation centers. Clinicians rarely knew when to initiate education about skin cancer risks and prevention including timing and scope, and rarely demonstrated understanding of the importance of reminders for and repeated education of patients. (National Kidney Foundation 2006) The NKF supported standard, formal, well timed skin cancer prevention information and sending reminders to KTRs at the beginning of summer.

Aims:

1. To explore culturally sensitive use of terms describing ethnic cultural perceptions of sun burning, pigment darkening after sun exposure and description of skin color by the amount of photoprotective pigment in the skin.
2. To pilot test the internet-based sun protection brochure with English speaking KTRs representing 3 ethnic groups: White, Black and Hispanic.
3. To explore understanding of the importance of sun protection and the KTRs' confidence in their being able to practice sun protection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of kidney transplantation within the last 5 years
* Speaks English
* Can see to read
* Lives in the greater Chicago area and can attend a cognitive interview session
* 18-85 years old

Exclusion Criteria:

* Unable to speak English
* Cognitive impairment or neurologic disease
* Dementia or insufficient cognitive skills to follow instructions provided at a sixth grade language level
* Has had a skin cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Use of sun protection | 6 weeks
  Use of sun protection will be measured using 10 questions about what a person regularly does in summer during a warm sunny day and during a cloudy day regarding: 1) use of sunscreen; 2) wearing hat; 3) shirt with sleeves; 4) sunglasses; and 5) staying in the shade. The scores for these questions will be summed to derive a dichotomous measure of sun protection use (1= use of sun protection often or always; 0 otherwise).

SECONDARY OUTCOMES:
Level of sun burn or skin irritation from the sun | 6 weeks
  Three telephone interviews will be done on Mondays after at least 2 holiday weekends in which the weather is reported as sunny or partly sunny by the national weather service (Memorial Day, 4th of July and Labor Day) as well as one sunny non-holiday weekend. The KTR will be asked if they experienced a sunburn or skin irritation. The response will be dichotomous (yes/no).
Forearm skin pigment | 6 weeks
  Skin pigment as measured by reflectance spectrophotometry, ranging from limited [225 area-under-the-curve (AUIC)] to dense (75 AUIC).

CONTACTS AND LOCATIONS:
Overall Officials: June K. Robinson, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Faculty Foundation, Chicago, Illinois, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- [Derived] Robinson JK, Friedewald JJ, Desai A, Gordon EJ. Response Across the Health-Literacy Spectrum of Kidney Transplant Recipients to a Sun-Protection Education Program Delivered on Tablet Computers: Randomized Controlled Trial. JMIR Cancer. 2015 Aug 18;1(2):e8. doi: 10.2196/cancer.4787. PMID 28410176
- [Derived] Robinson JK, Guevara Y, Gaber R, Clayman ML, Kwasny MJ, Friedewald JJ, Gordon EJ. Efficacy of a sun protection workbook for kidney transplant recipients: a randomized controlled trial of a culturally sensitive educational intervention. Am J Transplant. 2014 Dec;14(12):2821-9. doi: 10.1111/ajt.12932. Epub 2014 Nov 13. PMID 25395386
- [Derived] Guevara Y, Gaber R, Clayman ML, Gordon EJ, Friedewald J, Robinson JK. Sun protection education for diverse audiences: need for skin cancer pictures. J Cancer Educ. 2015 Mar;30(1):187-9. doi: 10.1007/s13187-014-0661-7. PMID 24788983